CLINICAL TRIAL: NCT01490008
Title: An Open-label, Single-center Triqal to Evaluate Systemic Exposure of Catechins From Commercially Available, Topically Applied Veregen 15% Ointment in Patients With External Anogenital Warts and From Oral Intake of Green Tea Beverage in Healthy Volunteers
Brief Title: Systemic Exposure of Catechins From Veregen 15% Ointment in Patients With External Anogenital Warts and From Oral Intake of Green Tea Beverage in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MediGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT 1023; 2011-004857-20 (EudraCT Number)
Record Dates: First submitted 2011-12-02; First posted 2011-12-12 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Anogenital Warts
MeSH Terms: conditions — Condylomata Acuminata | interventions — green tea extract polyphenone E; Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Veregen (Experimental): Veregen® (sinecatechins) Ointment, 15%, local application of 250 mg corresponding to 0.5 cm strand of ointment, 3 times daily (total dose of 750 mg/d)
  Interventions: Drug: Veregen
- Tea (Active Comparator): "Lipton® Green Limone", a green tea beverage; oral intake of 500 mL green tea, 3 times daily (total dose on 1500 mL/d)
  Interventions: Other: Green Tea

INTERVENTIONS:
Drug: Veregen — Patients in treatment arm 1 will apply Veregen® 15% ointment (approved commercial source in US) in a total of 750 mg/day for one week, corresponding to application of maximal about 106,9 mg catechins/d, thereof maximal 81 mg ECGg per day). Patients will be instructed to apply fix portions of 250 mg three times daily on the defined anogenital administration area.
  Arms: Veregen
Other: Green Tea — Healthy volunteers in treatment arm 2 will drink "Lipton® Green Limone" in a total of 1500 mL/d for one week, in portions of 500 mL three times daily after the meals
  Arms: Tea

SUMMARY:
Investigation of systemic catechin exposure following topically administered Veregen® 15% ointment in patients with external genital and perianal warts and following oral intake of a standardized green tea beverage in healthy subjects.

Pharmacokinetic parameters for the main catechin EGCg used as a marker of overall catechin exposure following dermal administration in the patient group will only be calculated if sufficiently consistent data can be obtained e.g. sufficient plasma catechin concentrations to pharmacokinetically evaluate plasma profiles for plasma catechin concentrations.

If applicable, a safety margin for ointment use might need to be established with respect to intolerable systemic exposures of catechins following application of Veregen® ointment.

In treatment arm 1, patients with anogenital warts will apply Veregen® 15% ointment 250 mg three times daily: in the morning, at midday, and in the evening on the defined anogenital administration area (total dose of 750 mg/d) for one week .

In treatment arm 2, healthy subjects will ingest 500 mL commercially available green tea beverage ("Lipton® Green Limone" distributed by PepsiCo Deutschland GmbH, Neu-Isenburg, Germany), three times daily in the morning, at midday, and in the evening (total dose of 1500 mL/d) for one week.

Plasma samples will be collected to aim for a complete pharmacokinetic assessment (over 24 hours) on Days 1 and 2 at Visit 2 and on Days 7 and 8 at Visit 3 (one week after first dosing).

To avoid any influence on overall systemic catechin exposure deriving from any other source than Veregen® or Lipton Green Tea, all subjects participating in the trial (patients and healthy volunteers) will be asked to follow a defined diet abstaining from food or beverages known to containing catechins (a list of all prohibited and allowed foods and beverages will be provided to all subjects).

For concomitant medication, only paracetamol and oral contraceptives are allowed.

ELIGIBILITY:
Inclusion Criteria:

For both subject groups (treatment arms 1 + 2):

1. Male and female subjects, 18 years of age or older at the time of enrollment. Subjects will be stratified by gender.
2. Written informed consent.
3. Ability to comply with the requirements of the study.
4. For male patients and partners of male patients who are of child-bearing potential: use of two methods of effective contraception (oral contraceptives, hormone containing intrauterine device, depot injection, hormone implant or sterilization plus condom during the treatment period is mandatory.
5. For women a negative pregnancy test and the willingness to use two methods of effective contraception (oral contraceptives, hormone containing intrauterine device, depot injection, hormone implant or sterilization plus condom during the treatment period is mandatory.

   For patients (treatment arm 1, additionally):
6. Clinical diagnosis of external genital and perianal warts which can be located: in men: over the glans penis, foreskin, penis shaft, and scrotum; in women: on the vulva; in both gender: in the inguinal, perineal, and perianal areas
7. For women a negative pregnancy test and willingness to abstain from cohabitation during the treatment phase.
8. For male patients willingness to abstain from cohabitation during the treatment phase.

   Exclusion Criteria:

   For both subject groups (treatment arms 1 + 2):
9. Participation in an investigational trial within 30 days prior to enrollment and for the whole study duration
10. Any current uncontrolled infection
11. Current known acute or chronic infection with Hepatitis virus B or C
12. Known Human immunodeficiency virus infection
13. Subjects with known history of instable diseases (diabetes, hypertension, etc.), severe gastritis or consuming diseases (cancer, multiple sclerosis, etc.), or liver or renal insufficiency.
14. Any chronic or acute condition including the skin, susceptible, in the opinion of the investigator, of interfering with the evaluation of the drug effect
15. Subject with any of the following:

    * quantitative hematology values deviating more than 20% of upper or lower normal values
    * clinical chemistry except electrolytes and liver enzymes deviating more than 50% of upper or lower normal values
    * liver enzymes exceeding twice the upper limit of normal range (ULN)
    * serum electrolytes deviating more than 20% of upper or lower normal values
    * abnormal results in urine supported by clinical evidence
    * laboratory values out of normal range and showing corresponding clinical signs or symptoms
16. Systemic intake of virostatics within 30 days prior to enrollment and for the whole study duration, with the exception of acyclovir and the related drugs famcyclovir and valcyclovir
17. Systemic intake of immunosuppressive or immunomodulatory medication or vaccination within 30 days prior to enrollment and for the whole study duration
18. Organ allograft recipient
19. Medication intake, including over the counter products and dietary supplements such as iodine, fluoride, or vitamins, which would interfere with study results, except paracetamol and oral contraceptives, within one week before and during the study course
20. Subjects not willing to avoid the consumption of food or beverage containing catechins, e.g. green, black or Oolong tea, red wine
21. For female patients: pregnancy or lactation
22. Blood transfusion within 30 days prior to enrollment
23. Subjects who are placed in an institution due to a judicial or official directive For patients (treatment arm 1; additionally)
24. Previous participation in a trial investigating sinecatechins in the treatment of external genital and perianal warts
25. Treatment of external genital warts within 14 days prior to enrollment and for the whole study duration
26. Current infection with Herpes genitalis or history of Herpes genitalis infection within the last 3 months prior to enrollment
27. Any current and/or recurrent pathologically relevant genital infections other than genital warts
28. Known allergies against any of the ingredients of the ointment
29. Internal (vaginal, urethral, or rectal) warts requiring treatment For healthy volunteers (treatment arm 2, additionally)
30. Known hereditary fructose intolerance, glucose-galactose malabsorption or saccharase-isomaltase deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Systemic exposure of green tea catechin EGC | At time points 0, i.e. prior to the morning ingestion of 500 mL of commercial green tea beverage or the morning application of 250 mg Veregen® 15%, and 0.5, 1, 2, 4, 6, 8, 10, 12, 14, and 24 hours afterwards.
  The primary objective of this trial is to investigate the systemic exposure, and, if possible, the plasma concentrations and pharmacokinetics of green tea catechin EGCg after topically applied Veregen® 15% ointment in patients with external genital warts and that following oral intake of commercially available green tea beverage by healthy subjects.
  On the sampling Days 1/2 and 7/8, blood samples of 3 mL each will be collected (non-fasting condition) at specified time points (see above)

CONTACTS AND LOCATIONS:
Locations (1):
- CardioSec Clinical Reasearch GmbH, Erfurt, Germany